CLINICAL TRIAL: NCT05547009
Title: A Randomized Trial Comparing Blended Learning Versus Face-to-face Learning in Cardiac Physiotherapy Students
Brief Title: Blended Learning Versus Face-to-face Learning in Cardiac Physiotherapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Elena Marques-Sule, Assistant Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IE1576047
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Learning; Students

STUDY DESIGN:
Intervention Model Description: An assessor-blinded two-armed randomized trial
Who Masked: Outcomes Assessor
Masking Description: The assessor was blinded to the participants interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blended-learning group (Experimental): The BL program included paced, asynchronous online learning modules and scheduled online activities with strategic face-to-face lectures.
  Interventions: Other: Blended-learning group
- Face-to-face learning group (Active Comparator): Face-to-face classes.
  Interventions: Other: Face-to-face learning group

INTERVENTIONS:
Other: Blended-learning group — The BL program included paced, asynchronous online learning modules and scheduled online activities with strategic face-to-face lectures. Resources: 1) Moodle platform: it was used as a virtual communication platform. 2) Online syllabus: an online specific syllabus about cardiac physiotherapy was developed. 3) Online glossary: an online glossary performed by the teacher was available for the students. 4) Online videos: several videos of international and national scientific societies were provided. 5) Websites: several links to websites of international and national scientific societies such as the European Society of Cardiology, the American Heart Association or the World Heart Federation were used. 6) Online activities: five four-question online activities were created. 7) Apps, using the app Ariadna to prevent from cardiovascular risk and look for defibrillators around; 8) Online tutorship, through an online communication platform (Blackboard Collaborate).
  Arms: Blended-learning group
Other: Face-to-face learning group — The FLG included: 1) Face-to-face classes; 2) Hardcopy syllabus; 3) Hardcopy scien-tific societies information; 4) Face-to-face activities: four questions per each theme; 5) Hardcopy glossary; and 6) Face-to-face tutorships. In all cases, the content of the infor-mation provided was the same as the information provided to the BLG, although in a face-to-face design.
  Arms: Face-to-face learning group

SUMMARY:
Blended learning (BL) combines both face-to-face learning (FL) and online learning. There is no evidence about the effects of a BL program in cardiac physiotherapy education. This study aimed at comparing the effectiveness of a BL program versus a FL program in Physiotherapy Degree students on knowledge, competencies, satisfaction, perceptions, usability, BL acceptance, attitudes and behaviours. An assessor-blinded randomized trial was performed.

DETAILED DESCRIPTION:
Blended learning (BL) combines both face-to-face learning (FL) and online learning. There is no evidence about the effects of a BL program in cardiac physiotherapy education. This study aimed at comparing the effectiveness of a BL program versus a FL program in Physiotherapy Degree students on knowledge, competencies, satisfaction, perceptions, usability, BL acceptance, attitudes and behaviours. An assessor-blinded randomized trial was performed. A total of 100 students were randomly allocated to a BL group (BLG, n=48), or a FL group (FLG, n=52). The BLG received face-to-face classes plus online re-sources (online syllabus, Moodle, scientific-based videos and websites, activities, glossary, and apps). The FLG received face-to-face classes and hardcopy resources (hardcopy syl-labus, scientific-based information, activities, and glossary). Knowledge, ethical and gen-der competencies, satisfaction, and perceptions were assessed pre- and post-intervention. Usability, BL acceptance, attitudes and behaviours were assessed post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being a student of Degree in Physiotherapy at the University of Valencia.
* Willing to participate

Exclusion Criteria:

* Previous cardiac physiotherapy training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Knowledge acquisition | 5 minutes
  Multiple-choice test. Score from 0 to 10 .The higher the score, the greater the knowledge.

SECONDARY OUTCOMES:
Cross-curricular ethical and gender competencies | 5 minute
  Higher Education, Transversal Skills and Gender Questionnaire. From 1 to 42. The higher the score, the more ethical and gender competencies are acquired.
Satisfaction with the program | 5 minute
  6-item Yang's Satisfaction Questionnaire. From 1 to 24. The higher the score, the greater the satisfaction with the program.
Perceptions and evaluation of the program | 5 minutes
  8-item Kavadella's Perceptions Questionnaire. From 1 to 40 points. The higher the score, the better the perceptions and evaluation of the program.
Usability of the virtual platform | 5 minutes
  System Usability Scale. The total SUS score (0 to 100) can be interpreted as not acceptable (0-64), acceptable (65 to 84), or excellent (85 to 100)
Blended-learning acceptance | 5 minutes
  4-item Blended Learning Acceptance Scale. From 1 to 28 points. The higher the score, the greater the acceptance.
Students' attitudes towards e-learning and e-learning behaviour | 5 minutes
  Questionnaire comprising 3 items (how much Moodle helped you, willingness of using Moodle, interest in e-learning). The higher score, the greater attitudes towards e-learning and e-learning behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Marqués Sulé, Dra, Principal Investigator — Univeristy of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

REFERENCES:
- [Background] Ng L, Seow KC, MacDonald L, Correia C, Reubenson A, Gardner P, Spence AL, Bunzli S, De Oliveira BIR. eLearning in Physical Therapy: Lessons Learned From Transitioning a Professional Education Program to Full eLearning During the COVID-19 Pandemic. Phys Ther. 2021 Apr 4;101(4):pzab082. doi: 10.1093/ptj/pzab082. PMID 33751113
- See also: Blended Learning: The impact of blackboard formative assessment on the final marks and students' perception of its effectiveness — https://pubmed.ncbi.nlm.nih.gov/32292428/
- See also: Blended learning in health education: three case studies — https://pubmed.ncbi.nlm.nih.gov/24458338/